CLINICAL TRIAL: NCT03135418
Title: Effect of Immersive Virtual Reality Usage on Upper Extremity Function in Stroke Patients: A Prospective, Double Blinded, Randomized Controlled Clinical Trial
Brief Title: Effect of Immersive Virtual Reality Usage on Upper Extremity Function in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AbantIBU-Neu1
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Stroke; Rehabilitation
Keywords: Virtual Reality
MeSH Terms: conditions — Stroke | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Patients' information and contact will be obtaioned from neurologist and willing participant's gender, age and stroke onset data will be processed with a random number generator. Patients will divide into two groups as intervention and control with a normal distrubution of gender, age and stroke onset.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both group will recevie conventional stroke rehabilitation. Intervention group will receive a Oculus Rift+Leap motion tracking supported upper extremity activities and control group will receive a sham virtual reality on focusing visual scenes without interaction.
  Outcomes will be recorded by physical therapist using SPSS and groups would not be specified with letter. Statistical analysis will be conducted by another researcher who does not aware of groups given numbers on SPSS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 25 stroke patients between the ages of 18-80, stroke duration of less than 2 months and not more than 2 years whose MMSE scores equal or above the 25 will be included in this study. Oculus Rift and Leap motion will be used to create an immersive interactive environment. Modified Ashworth Scale (MAS), Functional independence scale, self-care questionnaire,Action Research Arm Test, Fugl meyer upper extremity motor evaluations will be applied just before the rehabilitation program, after the application and at the end of 6 weeks.
  Interventions: Device: Intervention
- Control (Sham Comparator): 25 stroke patients between the ages of 18-80, stroke duration of less than 2 months and not more than 2 years whose MMSE scores equal or above the 25 will be included in this study. Oculus Rift a will be used to create an immersive visual environment.Patient will be watching the premade scenarios without interaction. Modified Ashworth Scale (MAS), Functional independence scale, self-care questionnaire, Action Research Arm Test, Fugl meyer upper extremity motor evaluations will be applied just before the rehabilitation program, after the application and at the end of 6 weeks.
  Interventions: Device: Control

INTERVENTIONS:
Device: Intervention — Patients will use virtual reality d4evice to play task oriented games like bowling, arrow shooting and home activity simulations which focuses upper extremity abduction, flexion and rotation movements. Each session will be a total of 45 minutes divided to 3 15 minute games. Sessions will held for 6 weeks each monday, wednesday and friday at same time for each patient.
  In addition to the virtual reality treatment program conventional rehabilitation therapies including neurodevelopmental facilitation techniques, physiotherapy, and occupational therapy and, where necessary, speech therapy will be applied according to the needs of the patient.
  Arms: Intervention
Device: Control — The control group will be included in the virtual reality program only focusing on visual scenes without upper extremity interaction. Bobath therapy, walking exercises, upper extremity active exercises, proprioceptive neuromuscular facial techniques will be applied to the control group for 6 weeks.
  Arms: Control

SUMMARY:
In this study we aimed to determine whether the additional rehabilitation with 3D virtual reality headsets provide any functional contribution to conventional rehabilitation techniques of upper extremity in patient with stroke.

Forty patients with stroke history no more than 2 years will be included in this study. Patients will randomly be divided into 2 groups as control and intervention. Conventional rehabilitation techniques will be applied for 4 weeks in both groups. Intervention group will receive a 3D virtual reality rehabilitation training, each lasts 45 minutes, with a special headset 3 times a week for 4 weeks in addition to conventional rehabilitation. Patients will be assessed with Fugl-Meyer, Action Research Arm Test and Functional Independence Measurement at baseline and 4 weeks after first assessment. It will be evaluated that whether 3d virtual reality rehabilitation training provides any benefit to stroke rehabilitation.

DETAILED DESCRIPTION:
According to the World Health Organization, cerebrovascular accident (CVA) or stroke is a rapidly evolving clinical manifestation, resulting death or lasting longer than 24 hours, due to local or general impairment of cerebral function without any cause other than vascular causes. These findings are due to the rapid loss of brain functions and impaired blood flow of the brain. Stroke is a cause of death and permanent neurological damage. After the disruption of the blood flow, the affected area of the brain loses its function. Hemiparesis and hemiplegia, aphasia, apraxia, dysarthria, loss of a visual field, and personality changes can occur. Stroke is a common neurological problem and one of the major causes of disability and death. In patients with stroke, the mortality rate is at the 30% level and there is an increasing the rate of morbidity. Therefore, stroke is one of the main causes of increasing health care costs in the adulthood. It has been shown that post-stroke rehabilitation might be effective in improving stroke symptoms and increasing independency however more study is needed to understand its specific effects.

Virtual reality applications are used predominantly in simulations and games, which has been developing rapidly with the development of day to day technology from 1980's. In medical field, it used for training of many diagnostic and therapeutic interventions such as laparoscopy and bronchoscopy in addition to rehabilitation. Reality and interactive video games have started to be used as a new treatment method in stroke rehabilitation. The advantage of this technology is that the types of activity which cannot be achieved or cannot be used in the clinical setting allow the patient to use it with abundant repetitive and visual feedback. Moreover, virtual reality programs are designed to be more fun and sustainable than traditional treatment programs. There is not any virtual reality device specially designed for use in therapy, but the game consoles used in the market can be modified and used for this purpose.

Oculus rift is an immersive console with the ability to create a real virtual environment. In a world where the individual is completely isolated from the outside and will be 360 degrees interactive in the designed environment, person has a near-real experience by seeing its own avatar and interacting with objects. There are two screens that are placed separately for each eye. These screens create stereoscopic 3D images by creating two separate images for the right and left eye. The accelerometer, gyroscope and magnetometer on the device are able to detect the direction and speed of movement. The greatest advantage of the oculus rift compared to other devices is that it prevents motion sickness such as nausea, dizziness and headache. Compared to older models, the new technology allows for a near-realistic environment design and object tracking, allowing the individual to use the device for extended periods of time without exposure to nausea and headaches.

Leap motion tracking system can mounted to oculus headset and it tracks the hands motion without requiring any other sensory device on the hand. Real time motion tracking provides a reliable visual output. Patients can interact virtual environment get feedbacks from program and see the result of their actions which is most needed to facilitate the plasticity. In order to get a good plasticity response 3 stimulation methods needed which is action from effected side, motor imagery and action observation. All 3 components can be achieved with usage of immersive virtual reality combined with a motion tracking.

Considering an 80% test power and an α > of 0.05, a minimum of 21 patients were needed for each group. Patients met the inclusion criteria will divide into two groups with a random number generator (considering gender, age and affected side) software as intervention and control groups.

At the first evaluation session, information of the cases that are considered appropriate to participate to the study will be recorded on the patient evaluation form. The assessments will be repeated at the beginning of the treatment schedule and at the end of the 4th week. Medical records like stroke onset, effected brain region, medications and detailed history will be provided by a neurologist.

The initial assessment will be done in the first day of the application before beginning the therapy and the last assessment will be done at the end of the 4th week. Mini Mental State Examination (MMSE) will be done to evaluate the cognitive status and cooperative skills. Patients scored 25 or more MMSE will be included to sudy.Modified Ashworth Scale (MAS), Functional independence scale, self-care questionnaire,Action Research Arm Test, Fugl meyer upper extremity motor evaluations will be applied before the rehabilitation program, after the intervention and at the end of 4 weeks.

It is considered that the use of oculus rift device in rehabilitation; i) may increase the efficiency of stroke rehabilitation and functional independence by increasing the participation of individuals ii) may increase the perception of the correct movement of the individuals iii) may allow measuring the effectiveness of rehabilitation numerically, different from other subjective methods.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate
* Mini-Mental State Test score equal or above 25
* Modified Ashworth Scale Score lover then 3

Exclusion Criteria:

* Secondary neurological diseases
* Recurrent strokes
* Reduced or lost visual field on both or single eye(s)
* Full paralysis on affected side

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-06 (Actual)

PRIMARY OUTCOMES:
Fugl meyer upper extremity motor evaluations | 6 weeks
  Evaluates and measures recovery in post-stroke hemiplegic patients. Motor Test requires Tennis ball, A small spherical shaped container, A tool to administer reflex tests, Enough space is needed for a patient to move around freely, if possible space should be a quiet

SECONDARY OUTCOMES:
Functional independence scale | 6 weeks
  Measures the level of a patient's disability and indicates how much assistance is needed for the individual to carry out activities of daily living
Performance Assessment of Self-Care Skills (PASS) | 6 weeks
  Purpose of PASS is to demonstrate independence, adequacy, and safety are rated on four-point scales.
Action Research Arm Test (ARAT) | 6 weeks
  Assesses upper limb functioning using observational methods. Focuses on grip, grasp and pinch motions of hand

CONTACTS AND LOCATIONS:
Overall Officials: Şule Aydın Türkoğlu, M.D., Principal Investigator — Abant Izzet Baysal University; Ramazan Kurul, Ms.C, Principal Investigator — Abant Izzet Baysal University; Muhammed Nur Öğün, M.D., Study Director — Abant Izzet Baysal University; Şebnem Avcı, Ph.D., Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
After publication of article all outcomes will be open to others researches with an excel data sheet. Researchers can contact corresponding researcher with his contact mail and request data.